CLINICAL TRIAL: NCT04714125
Title: Prognostic Value of Flow-mediated Dilation in Hospitalized Patients With SARS-CoV-2 Infection: an Observational Prospective Study
Brief Title: Prognostic Value of Flow-mediated Dilation in Hospitalized COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FMDCOVID
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: endothelial function; flow-mediated dilation; vascular function; carotid intima-media thickness
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with COVID-19: Patients hospitalized with COVID-19 from the General Hospital of the University of Sao Paulo, Brazil.

SUMMARY:
This study will evaluate the associations between vascular parameters and clinical outcomes in patients hospitalized with COVID-19.

The vascular function and structure of individuals with COVID-19 admitted to the General Hospital of the University of Sao Paulo will be assessed in the first 72 hours of hospitalization. Then, participants will be followed up until hospital discharge/death.

Logistical regressions will be run to evaluate if vascular function/structure can predict ICU admissions, intubation, thrombosis or death.

DETAILED DESCRIPTION:
This is a prospective cohort study conducted at the General Hospital of the University of São Paulo Medical School (HCFMUSP). Male and female participants with SARS-CoV-2 and recently admitted to the hospital (≤ 72 hours) will be recruited at the emergency department and outpatient clinics at the HCFMUSP. Immediately upon recruitment, participants will perform the assessment of flow mediated dilation of the brachial artery and the assessment of carotid intima-media thickness. Subsequently, they will be followed during the entire period of hospitalization.

The present study will employ as primary endpoint a composite of ICU admission, intubation or mortality during the period of hospitalization. Cardiovascular complications, such as arterial (AE), deep venous (DVP) or pulmonary embolism (PE) , acute myocardial infarction (AMI), stroke, cardiac arrest, atrial fibrillation and acute kidney injury will be considered secondary endpoints.

The association between the vascular parameters and clinical outcomes will be examined by a multivariate logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with SARS-CoV-2
* Recently admitted to the hospital (≤ 72 hours)
* Not yet proceeded to ICU care

Exclusion Criteria:

* Patients transferred from other hospitals
* Participants in delirium state
* Participants with a recent history of endotracheal intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adults with SARS-CoV-2 and recently admitted (≤ 72 hours) to the General Hospital of the Faculty of Medicine of the University of Sao Paulo.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome | Up to hospital discharge, an average of 4 weeks
  A composite outcome including ICU admission, intubation and all-cause mortality

SECONDARY OUTCOMES:
All-cause mortality | Up to hospital discharge, an average of 4 weeks
  All-cause mortality rate along the study
ICU admission | Up to hospital discharge, an average of 4 weeks
  Admission to the ICU along the study
Intubation | Up to hospital discharge, an average of 4 weeks
  Necessity of intubation along the study
Cardiovascular complications | Up to hospital discharge, an average of 4 weeks
  Cardiovascular complications, such as arterial, deep venous or pulmonary embolism, acute myocardial infarction, stroke, cardiac arrest, atrial fibrillation and acute kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da USP - HCFMUSP, São Paulo, Brazil